CLINICAL TRIAL: NCT04741971
Title: Whether Probiotics Use in Neonate and Infant Improve Their Mother's Life Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chao Hsiao, Co-Principal Investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P00001711
Record Dates: First submitted 2021-01-12; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Postpartum Depression; Quality of Life; Functional Gastrointestinal Disorders; Probiotics
Keywords: Postpartum Depression; Probiotics; infantile colic
MeSH Terms: conditions — Depression, Postpartum; Gastrointestinal Diseases; Colic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): Will give Probiotics with Vit.D 3
  Interventions: Dietary Supplement: Probiotics group
- Non-probiotics group (Placebo Comparator): Will give Vit. D3 as placebo
  Interventions: Dietary Supplement: Non-probiotics group

INTERVENTIONS:
Dietary Supplement: Probiotics group — Will give Probiotics with Vitamin D3 one drop per day for 90 days
  Arms: Probiotics group
Dietary Supplement: Non-probiotics group — Will give Vitamin D3 five drops per day for 90 days
  Arms: Non-probiotics group

SUMMARY:
Postpartum depression and poor quality of life during postpartum were an vital issue in recent years. Infant's health condition was thought to be a possible reasons related mother's postpartum quality of life, and functional gastrointestinal disorders such as infantile colic and regurgitation were common problem during infant period. Previous study revealed that probiotics may improve the infant's discomfort caused by functional gastrointestinal disorders. Thus, this study aimed to investigate whether probiotics use in neonate and infant improve their mother's life quality?

DETAILED DESCRIPTION:
This is single blinded intervention study. The investigators will invite mother to participate in the project after giving birth. At week 0, mother who meet the eligibility criteria will be randomized in a single-blind study in a 1:1 ratio to probiotics with Vit. D3 (five drops per day) or Vit. D3 (placebo) (single drop per day) for 90 days. The follow-up will be at the 1, 3 and 6 months all the subjects.

ELIGIBILITY:
<Participants of neonates>

Inclusion Criteria :

* Gestational age more than 37 to less than 41 weeks
* Age less than 1 week on entry into the study
* Birth weight adequate for gestational age
* Apgar score of more than 8 at 10 minutes

Exclusion Criteria:

* Congenital disorders and/or clinical or physical alterations at clinical examination
* Antibiotic or probiotic administration before inclusion
* Admission to ICU

<Participants of neonates' mother>

Inclusion Criteria:

* Aged between 20-50 and baby included in our study

Exclusion Criteria:

* Diagnosed as psychiatric disease during antepartum period or before pregnancy

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-02-18 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Sleep Quality | at their child birth
  Maternal Sleep Quality assessed by the Pittsburgh Sleep Quality Index (PSQI): a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. In scoring the PSQI, there are seven component scores with each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce total score (range 0 to 21). Higher scores indicate worse sleep quality.
Maternal Sleep Quality | at their child 1-month-old
  Maternal Sleep Quality assessed by the Pittsburgh Sleep Quality Index (PSQI): a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. In scoring the PSQI, there are seven component scores with each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce total score (range 0 to 21). Higher scores indicate worse sleep quality.
Maternal Sleep Quality | at their child 3-month-old
  Maternal Sleep Quality assessed by the Pittsburgh Sleep Quality Index (PSQI): a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. In scoring the PSQI, there are seven component scores with each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce total score (range 0 to 21). Higher scores indicate worse sleep quality.
Maternal Sleep Quality | at their child 6-month-old
  Maternal Sleep Quality assessed by the Pittsburgh Sleep Quality Index (PSQI): a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. In scoring the PSQI, there are seven component scores with each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce total score (range 0 to 21). Higher scores indicate worse sleep quality.
Maternal quality of life | at their child birth
  Maternal quality of life assessed by World Health Organization Quality of Life (WHOQOL) questionnaire - Brief, Taiwan version: a questionnaire including 28 items with each score 0-4. Higher score indicate better quality of life.
Maternal quality of life | at their child 1-month-old
  Maternal quality of life assessed by World Health Organization Quality of Life (WHOQOL) questionnaire - Brief, Taiwan version: a questionnaire including 28 items with each score 0-4. Higher score indicate better quality of life.
Maternal quality of life | at their child 3-month-old
  Maternal quality of life assessed by World Health Organization Quality of Life (WHOQOL) questionnaire - Brief, Taiwan version: a questionnaire including 28 items with each score 0-4. Higher score indicate better quality of life.
Maternal quality of life | at their child 6-month-old
  Maternal quality of life assessed by World Health Organization Quality of Life (WHOQOL) questionnaire - Brief, Taiwan version: a questionnaire including 28 items with each score 0-4. Higher score indicate better quality of life.
Maternal risk of postnatal depression | at their child birth
  Maternal risk of postnatal depression assessed by Edinburgh Postnatal Depression Scale: a set of 10 screening questions with each score 0 to 3 that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. Higher score indicate higher risk of postnatal depression.
Maternal risk of postnatal depression | at their child birth 1-month-old
  Maternal risk of postnatal depression assessed by Edinburgh Postnatal Depression Scale: a set of 10 screening questions with each score 0 to 3 that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. Higher score indicate higher risk of postnatal depression.
Maternal risk of postnatal depression | at their child birth 3-month-old
  Maternal risk of postnatal depression assessed by Edinburgh Postnatal Depression Scale: a set of 10 screening questions with each score 0 to 3 that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. Higher score indicate higher risk of postnatal depression.
Maternal risk of postnatal depression | at their child birth 6-month-old
  Maternal risk of postnatal depression assessed by Edinburgh Postnatal Depression Scale: a set of 10 screening questions with each score 0 to 3 that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. Higher score indicate higher risk of postnatal depression.

SECONDARY OUTCOMES:
Neonate and infant' condition of functional gastrointestinal disorders | at baby's 1-month-old
  Neonate and infant' condition of functional gastrointestinal disorders including infantile colic and regurgitation assessed by the questionnaires according to ROME-IV criteria, and higher score indicate worse condition of functional gastrointestinal disorders in infancy.
Neonate and infant' condition of functional gastrointestinal disorders | at baby's 3-month-old
  Neonate and infant' condition of functional gastrointestinal disorders including infantile colic and regurgitation assessed by the questionnaires according to ROME-IV criteria, and higher score indicate worse condition of functional gastrointestinal disorders in infancy.
Neonate and infant' condition of functional gastrointestinal disorders | at baby's 6-month-old
  Neonate and infant' condition of functional gastrointestinal disorders including infantile colic and regurgitation assessed by the questionnaires according to ROME-IV criteria, and higher score indicate worse condition of functional gastrointestinal disorders in infancy.
Neonate and infant' diaper dermatitis | at baby's 1-month-old
  Neonate and infant' diaper dermatitis assessed by the self-rated questionnaire to determine the condition of diaper dermatitis.
Neonate and infant' diaper dermatitis | at baby's 3-month-old
  Neonate and infant' diaper dermatitis assessed by the self-rated questionnaire to determine the condition of diaper dermatitis.
Neonate and infant' diaper dermatitis | at baby's 6-month-old
  Neonate and infant' diaper dermatitis assessed by the self-rated questionnaire to determine the condition of diaper dermatitis.
Neonate and infant' atopic dermatitis | at baby's 1-month-old
  Neonate and infant' atopic dermatitis assessed by the self-rated questionnaire to determine the condition of atopic dermatitis
Neonate and infant' atopic dermatitis | at baby's 3-month-old
  Neonate and infant' atopic dermatitis assessed by the self-rated questionnaire to determine the condition of atopic dermatitis
Neonate and infant' atopic dermatitis | at baby's 6-month-old
  Neonate and infant' atopic dermatitis assessed by the self-rated questionnaire to determine the condition of atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsun Chang, Study Chair — Department of Pediatrics, Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation,Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Will share all IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: May be on December 2024
Access Criteria: Will be published

DOCUMENTS (1):
  • Study Protocol (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04741971/Prot_000.pdf